CLINICAL TRIAL: NCT03492372
Title: Molecular Characterization of Spinal Tissue
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, A. Noelle Larson, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 14-008177
Record Dates: First submitted 2018-01-25; First posted 2018-04-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Spinal tissues removed as discarded tissue, waste, or surgical debris. Examples: disc, cartilage, ligament
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Spine patients: Patients undergoing spine surgery where spinal tissue is discarded/removed will be recruited. Tissue samples will be used to look at normal and pathologic molecular signatures.
  Interventions: Other: Waste tissues are collected at the time of spinal surgery.

INTERVENTIONS:
Other: Waste tissues are collected at the time of spinal surgery. — This is a single visit study. Waste tissues are collected at the time of spinal surgery.

SUMMARY:
The researchers are trying to identify molecular mechanisms that control spine deformity and degenerative changes that can be used for therapeutic strategies.

DETAILED DESCRIPTION:
Discarded surgical material from spinal procedures is collected. RNA analysis and other tests on the tissue is performed to determine markers of pathologic disease and to develop pharmacologic treatment strategies for pediatric spinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults undergoing surgical procedures where spinal tissues are removed as a normal part of their procedure. Material from adults may be collected as a control group.

Exclusion Criteria:

* Surgeries where spinal tissues are not being removed.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing spinal surgery where spinal tissues (disc, cartilage, ligament, etc.) is removed as discarded tissue, waste, or surgical debris.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-03-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
RNA expression | Baseline
  Measure RNA levels in spinal tissues samples (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: A.Noelle Larson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No